CLINICAL TRIAL: NCT02749279
Title: Adherence to Lipid Lowering Therapy After Cardiac Rehabilitation (LLT-Rehabilitation-Registry)
Brief Title: Lipid Lowering Therapy After Cardiac Rehabilitation LLT-R-Registry
Acronym: LLT-R-Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Paracelsus Harz Clinic Bad Suderode. (Other)
Collaborators: KKS Netzwerk (Network)
Responsible Party: Sponsor
Other Study IDs: ParacelsusHCBS 01/16
Record Dates: First submitted 2016-04-08; First posted 2016-04-22 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-03

CONDITIONS: Lipid Lowering Therapy After Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The most important drugs for evidence based lipid lowering treatment (LLT) in CHD are statins. All patients with established CHD should be treated with statins irrespective of low density lipoprotein (LDL) cholesterol (LDL-C) levels. The goals of treatment are LDL-C below 1.8 mmol/L (70 mg/dL) or 50% LDL-C reduction when target level cannot be reached. Unfortunately, several patients cannot achieve treatment targets also related to the serious problem of adherence to therapy, which includes also LLT.

DETAILED DESCRIPTION:
In German rehabilitation clinics the number of patients who has a clear indication for LLT is continuously high since years. Approximately 2,000 patients with cardiac diseases were treated per year per clinic and momentarily approximately three fourth of them have an indication for LLT, mainly patients with CHD. The main length of stay in German rehabilitation clinics is 21 days, which gives the chance and the necessity to optimize LLT, since in approximately 50% of all patients with an indication for LLT treatment targets are not achieved.

After patients will give written informed consent, data will be collected. Here, all relevant baseline parameters (drug treatment, indication for rehabilitation, all clinical diagnoses, age, sex, BMI, echocardiographic parameters such as left ventricular ejection fraction, laboratory parameters corresponding to the recording standard of the clinic, etc.) will be recorded in a central database (online-CRF). Furthermore, as the main topic of interest of the study, LLT at baseline, LLT during the rehabilitation phase, and LLT treatment at discharge including the recommendation given for the home physicians regarding LLT in the discharge letter will be collected. Here, according to the AHA/ACC Guideline (9) LLT will be stratified in low-intensity statin therapy (Simvastatin 10mg, Pravastatin 10-20mg, Lovastatin 20mg, Fluvastatin 20-40mg), moderate-intensity statin therapy (Atorvastatin 10-20mg, Rosuvastatin 5-10mg, Simvastatin 20-40mg, Pravastatin 40-80mg, Lovastatin 40mg, Fluvastatin 80mg) and high-intensity statin therapy (Atorvastatin 40-80mg, Rosuvastatin 20-40mg). Furthermore, data on other lipid lowering drugs such as cholesterol resorption inhibitors, fibrates and PCSK-9 inhibitors will be collected. Adverse events related to drug therapy will be further collected and submitted to the German health authorities. Furthermore, serious adverse events (SAE), for drugs manufactured by Sanofi-Aventis, Zentiva or Genzyme, will be submitted to Sanofi-Aventis.

At discharge patient will receive a questionnaire, which includes questions about change of drug treatment during the next 12 months. Here, patients will record prospectively whether medication has been changed and if so, why, and who changed it.

After discharge patients will be contacted by mail after three and twelve months. Patients will asked in addition to the questionnaire at discharge about drug therapy with special regards to LLT Changes in medication will be documented by comparison of drug list at discharge with the patient reported drugs, which are taken at time of follow-up.

Furthermore, general questions about other drug therapy, re-hospitalizations especially in connection with atherosclerotic diseases such as cardiac death, Re-PCI, Bypass, pulmonary embolism, TIA/ stroke, bleeding, ACS/MI, and others are recorded. In this disease registry these endpoints will be recorded separately and statistically analyzed, however not defined as AE and not recorded as such. Patients will be further asked whether other adverse events occurred and whether they may be related to drug therapy. If AEs in relation to drug therapy will be reported these information will be submitted to the German health authorities. SAE, with drugs manufactured by Sanofi-Aventis,Zentiva or Genzyme will be submitted to Sanofi-Aventis.

Clinical research organization (CRO) will carry out

* GCP-compliant data management: eCRF - creation including validation and consistency checks, input and training regarding the manual (while auditors meeting), online delivery incl. license allocation and support, patient registration, query management, data export to biometrics.
* GCP-compliant quality control (Clinical Monitoring), setup process including monitoring, initiating the inspection once centrally (auditors meeting) including a total of 22 on-site visits (2 / center).
* Study preparation incl. review of study documents, submission to ethics committees, supporting the drafting and implementation, creation of test folder and the "Trial Master Files"
* Study Coordination and care of the on-site files

ELIGIBILITY:
Inclusion Criteria:

* Lipid lowering therapy after cardiac rehabilitation

Exclusion Criteria:

* Inability or refusal to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with CHD, who will be admitted for cardiac rehabilitation to the participating German rehabilitation clinics and in whom LLT is indicated will be included. Written informed consent will be obtained from each participant. Beginning of the study is 1st May 2016, the inclusion of the last patient is expected on 30th April 2016. Follow-up: at 3 and 12 months, respectively, inclusion of 100 participants per clinic is expected.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Data collection (Adherence to lipid lowering therapy after cardiac rehabilitation) | 12 Months
  Adherence to lipid lowering therapy after cardiac rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus Harz Clinic Bad Suderode, Quedlinburg, Saxony-Anhalt, Germany